CLINICAL TRIAL: NCT03930680
Title: Prevention of Heart Failure Induced by Doxorubicin With Early Administration of Dexrazoxane in Patients With Breast Cancer
Brief Title: Prevention of Heart Failure Induced by Doxorubicin With Early Administration of Dexrazoxane
Acronym: PHOENIX1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 262180; R01HL151993 (NIH)
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Degradation of Top2b and Top2a in Human by Dexrazoxane; Time Course and Degradation of Top2b in Human by Dexrazoxane; Effects of Dexrazoxane on Healthy Human
Keywords: Dexrazoxane; Topoisomerase 2b; Human; Doxorubicin cardio-toxicity; Cardio-oncology; Onco-cardiology; Prevention of cardio-toxicity by doxorubicin; Early administration of dexrazoxane
MeSH Terms: interventions — Dexrazoxane

STUDY DESIGN:
Intervention Model Description: Each subject will receive one dose of dexrazoxane.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Dexrazoxane 100mg/m2 (Experimental): one dose of 100mg/m2 dexrazoxane
  Interventions: Drug: Dexrazoxane
- Dexrazoxane 200mg/m2 (Experimental): one dose of 200mg/m2 dexrazoxane
  Interventions: Drug: Dexrazoxane
- Dexrazoxane 300mg/m2 (Experimental): one dose of 300mg/m2 dexrazoxane
  Interventions: Drug: Dexrazoxane
- Dexrazoxane 400mg/m2 (Experimental): one dose of 400mg/m2 dexrazoxane
  Interventions: Drug: Dexrazoxane
- Dexrazoxane 500mg/m2 (Experimental): one dose of 500 mg/m2
  Interventions: Drug: Dexrazoxane

INTERVENTIONS:
Drug: Dexrazoxane — One dose of dexrazoxane
  Other Names: Zinecard

SUMMARY:
The purpose of this research study is to determine whether early administration of Dexrazoxane prevents Doxorubicin induced cardiotoxicity.

DETAILED DESCRIPTION:
This is a study on volunteers to determine effective dose of dexrazoxane in degrading Topoisomerase 2 b in human blood samples. Each participant will receive one dose of dexrazoxane. Blood samples will be collected to determine the time course and degradation of Topoisomerase 2b and Topoisomerase 2a

ELIGIBILITY:
Inclusion Criteria:

* Women,
* Age 18-65,
* Not pregnant, Not currently breast feeding
* No current illness,

Exclusion Criteria:

* Pregnancy, currently breast feeding
* Current illness,
* History of cardiac, or renal disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2025-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ming Chang, MD,MPH, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang HM, Moudgil R, Scarabelli T, Okwuosa TM, Yeh ETH. Cardiovascular Complications of Cancer Therapy: Best Practices in Diagnosis, Prevention, and Management: Part 1. J Am Coll Cardiol. 2017 Nov 14;70(20):2536-2551. doi: 10.1016/j.jacc.2017.09.1096. PMID 29145954
- [Background] Zhang S, Liu X, Bawa-Khalfe T, Lu LS, Lyu YL, Liu LF, Yeh ET. Identification of the molecular basis of doxorubicin-induced cardiotoxicity. Nat Med. 2012 Nov;18(11):1639-42. doi: 10.1038/nm.2919. Epub 2012 Oct 28. PMID 23104132
- [Background] Lipshultz SE, Lipsitz SR, Kutok JL, Miller TL, Colan SD, Neuberg DS, Stevenson KE, Fleming MD, Sallan SE, Franco VI, Henkel JM, Asselin BL, Athale UH, Clavell LA, Michon B, Laverdiere C, Larsen E, Kelly KM, Silverman LB. Impact of hemochromatosis gene mutations on cardiac status in doxorubicin-treated survivors of childhood high-risk leukemia. Cancer. 2013 Oct 1;119(19):3555-62. doi: 10.1002/cncr.28256. Epub 2013 Jul 16. PMID 23861158
- [Background] Tewey KM, Rowe TC, Yang L, Halligan BD, Liu LF. Adriamycin-induced DNA damage mediated by mammalian DNA topoisomerase II. Science. 1984 Oct 26;226(4673):466-8. doi: 10.1126/science.6093249.
- [Background] Olson LE, Bedja D, Alvey SJ, Cardounel AJ, Gabrielson KL, Reeves RH. Protection from doxorubicin-induced cardiac toxicity in mice with a null allele of carbonyl reductase 1. Cancer Res. 2003 Oct 15;63(20):6602-6. PMID 14583452
- [Background] Azuma Y, Arnaoutov A, Dasso M. SUMO-2/3 regulates topoisomerase II in mitosis. J Cell Biol. 2003 Nov 10;163(3):477-87. doi: 10.1083/jcb.200304088. Epub 2003 Nov 3. PMID 14597774
- [Background] Lyu YL, Kerrigan JE, Lin CP, Azarova AM, Tsai YC, Ban Y, Liu LF. Topoisomerase IIbeta mediated DNA double-strand breaks: implications in doxorubicin cardiotoxicity and prevention by dexrazoxane. Cancer Res. 2007 Sep 15;67(18):8839-46. doi: 10.1158/0008-5472.CAN-07-1649. PMID 17875725
- [Background] Swain SM, Whaley FS, Gerber MC, Weisberg S, York M, Spicer D, Jones SE, Wadler S, Desai A, Vogel C, Speyer J, Mittelman A, Reddy S, Pendergrass K, Velez-Garcia E, Ewer MS, Bianchine JR, Gams RA. Cardioprotection with dexrazoxane for doxorubicin-containing therapy in advanced breast cancer. J Clin Oncol. 1997 Apr;15(4):1318-32. doi: 10.1200/JCO.1997.15.4.1318. PMID 9193323
- [Background] Bluethmann SM, Mariotto AB, Rowland JH. Anticipating the "Silver Tsunami": Prevalence Trajectories and Comorbidity Burden among Older Cancer Survivors in the United States. Cancer Epidemiol Biomarkers Prev. 2016 Jul;25(7):1029-36. doi: 10.1158/1055-9965.EPI-16-0133. PMID 27371756
- [Background] Chang HM, Okwuosa TM, Scarabelli T, Moudgil R, Yeh ETH. Cardiovascular Complications of Cancer Therapy: Best Practices in Diagnosis, Prevention, and Management: Part 2. J Am Coll Cardiol. 2017 Nov 14;70(20):2552-2565. doi: 10.1016/j.jacc.2017.09.1095. PMID 29145955
- [Background] Armstrong GT, Kawashima T, Leisenring W, Stratton K, Stovall M, Hudson MM, Sklar CA, Robison LL, Oeffinger KC. Aging and risk of severe, disabling, life-threatening, and fatal events in the childhood cancer survivor study. J Clin Oncol. 2014 Apr 20;32(12):1218-27. doi: 10.1200/JCO.2013.51.1055. Epub 2014 Mar 17. PMID 24638000
- [Background] Darby SC, Cutter DJ, Boerma M, Constine LS, Fajardo LF, Kodama K, Mabuchi K, Marks LB, Mettler FA, Pierce LJ, Trott KR, Yeh ET, Shore RE. Radiation-related heart disease: current knowledge and future prospects. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):656-65. doi: 10.1016/j.ijrobp.2009.09.064. PMID 20159360
- [Background] Swain SM, Vici P. The current and future role of dexrazoxane as a cardioprotectant in anthracycline treatment: expert panel review. J Cancer Res Clin Oncol. 2004 Jan;130(1):1-7. doi: 10.1007/s00432-003-0498-7. Epub 2003 Oct 17. PMID 14564513
- [Background] Yeh ET, Chang HM. Oncocardiology-Past, Present, and Future: A Review. JAMA Cardiol. 2016 Dec 1;1(9):1066-1072. doi: 10.1001/jamacardio.2016.2132. PMID 27541948
- [Background] Tan C, Tasaka H, Yu KP, Murphy ML, Karnofsky DA. Daunomycin, an antitumor antibiotic, in the treatment of neoplastic disease. Clinical evaluation with special reference to childhood leukemia. Cancer. 1967 Mar;20(3):333-53. doi: 10.1002/1097-0142(1967)20:33.0.co;2-k. No abstract available. PMID 4290058
- [Background] Von Hoff DD, Layard MW, Basa P, Davis HL Jr, Von Hoff AL, Rozencweig M, Muggia FM. Risk factors for doxorubicin-induced congestive heart failure. Ann Intern Med. 1979 Nov;91(5):710-7. doi: 10.7326/0003-4819-91-5-710. PMID 496103
- [Background] Doroshow JH. Effect of anthracycline antibiotics on oxygen radical formation in rat heart. Cancer Res. 1983 Feb;43(2):460-72. PMID 6293697
- [Background] Doroshow JH, Locker GY, Myers CE. Enzymatic defenses of the mouse heart against reactive oxygen metabolites: alterations produced by doxorubicin. J Clin Invest. 1980 Jan;65(1):128-35. doi: 10.1172/JCI109642. PMID 7350193
- [Background] Doroshow JH. Doxorubicin-induced cardiac toxicity. N Engl J Med. 1991 Mar 21;324(12):843-5. doi: 10.1056/NEJM199103213241210. No abstract available. PMID 1997858
- [Background] Gianni L, Herman EH, Lipshultz SE, Minotti G, Sarvazyan N, Sawyer DB. Anthracycline cardiotoxicity: from bench to bedside. J Clin Oncol. 2008 Aug 1;26(22):3777-84. doi: 10.1200/JCO.2007.14.9401. PMID 18669466
- [Background] Herman EH, Ferrans VJ, Myers CE, Van Vleet JF. Comparison of the effectiveness of (+/-)-1,2-bis(3,5-dioxopiperazinyl-1-yl)propane (ICRF-187) and N-acetylcysteine in preventing chronic doxorubicin cardiotoxicity in beagles. Cancer Res. 1985 Jan;45(1):276-81. PMID 3917371
- [Background] Myers C, Bonow R, Palmeri S, Jenkins J, Corden B, Locker G, Doroshow J, Epstein S. A randomized controlled trial assessing the prevention of doxorubicin cardiomyopathy by N-acetylcysteine. Semin Oncol. 1983 Mar;10(1 Suppl 1):53-5. No abstract available. PMID 6340204
- [Background] Martin E, Thougaard AV, Grauslund M, Jensen PB, Bjorkling F, Hasinoff BB, Tjornelund J, Sehested M, Jensen LH. Evaluation of the topoisomerase II-inactive bisdioxopiperazine ICRF-161 as a protectant against doxorubicin-induced cardiomyopathy. Toxicology. 2009 Jan 8;255(1-2):72-9. doi: 10.1016/j.tox.2008.10.011. Epub 2008 Oct 25. PMID 19010377
- [Background] Capranico G, Tinelli S, Austin CA, Fisher ML, Zunino F. Different patterns of gene expression of topoisomerase II isoforms in differentiated tissues during murine development. Biochim Biophys Acta. 1992 Aug 17;1132(1):43-8. doi: 10.1016/0167-4781(92)90050-a. PMID 1380833
- [Background] Wang J, Zhang S, Rabinovich B, Bidaut L, Soghomonyan S, Alauddin MM, Bankson JA, Shpall E, Willerson JT, Gelovani JG, Yeh ET. Human CD34+ cells in experimental myocardial infarction: long-term survival, sustained functional improvement, and mechanism of action. Circ Res. 2010 Jun 25;106(12):1904-11. doi: 10.1161/CIRCRESAHA.110.221762. Epub 2010 May 6. PMID 20448213
- [Background] Hasinoff BB. Chemistry of dexrazoxane and analogues. Semin Oncol. 1998 Aug;25(4 Suppl 10):3-9. PMID 9768817
- [Result] Chang HM, Hsu JY, Ahn C, Yeh ETH. Prevention of Heart Failure Induced by Doxorubicin with Early Administration of Dexrazoxane (PHOENIX Study): dose response and time course of dexrazoxane-induced degradation of topoisomerase 2b. Cardiooncology. 2025 May 2;11(1):42. doi: 10.1186/s40959-025-00339-0. PMID 40317097

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexrazoxane 100mg/m2 | Dexrazoxane 200mg/m2 | Dexrazoxane 300mg/m2 | Dexrazoxane 400mg/m2 | Dexrazoxane 500mg/m2
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexrazoxane 100mg/m2 | Dexrazoxane 200mg/m2 | Dexrazoxane 300mg/m2 | Dexrazoxane 400mg/m2 | Dexrazoxane 500mg/m2 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 5 | 5 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 5 | 5 | 25
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 0 | 0 | 3
  White | 4 | 3 | 3 | 5 | 4 | 19
  More than one race | 1 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 5 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Participants With 95% Reduction in Topoisomerase 2 b From Baseline
Description: Number of participants with 95% reduction in topoisomerase 2 b from baseline is reported in the Outcome Measure Data Table
Time Frame: 8 hours after dexrazoxane administration
Measure: Count of Participants; unit: Participants
Arm/Group | Dexrazoxane 100mg/m2 | Dexrazoxane 200mg/m2 | Dexrazoxane 300mg/m2 | Dexrazoxane 400mg/m2 | Dexrazoxane 500mg/m2
Number analyzed (Participants) | 4 | 5 | 5 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: The adverse event data were collected on the date of one dose dexrazoxane infusion, one day and two days after infusion, and one week after infusion. Some of the participants required a visit two weeks after one dose dexrazoxane infusion. Adverse event data were collected during the visit.
Arm/Group | Dexrazoxane 100mg/m2 | Dexrazoxane 200mg/m2 | Dexrazoxane 300mg/m2 | Dexrazoxane 400mg/m2 | Dexrazoxane 500mg/m2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 1/5 | 2/5 | 0/5 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexrazoxane 100mg/m2 (N=5) | Dexrazoxane 200mg/m2 (N=5) | Dexrazoxane 300mg/m2 (N=5) | Dexrazoxane 400mg/m2 (N=5) | Dexrazoxane 500mg/m2 (N=5)
bruising (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
pain (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
anemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 1
other (General disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
In animal studies, Top2b expression can be directly measured in heart tissues; however, this is not feasible in human participants. Therefore, peripheral blood mononuclear cells were chosen as a surrogate tissue to assess Top2b degradation. Our study participants were adult women, so the dose-response curve and time course may not be applicable to the pediatric cancer population. Our study evaluates the dose-response and time course of dexrazoxane's effects on Top2a and Top2b expression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT03930680/Prot_000.pdf
  • Informed Consent Form (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT03930680/ICF_001.pdf